CLINICAL TRIAL: NCT07288411
Title: Pilot Study of the Effects of Transcutaneous Non-Invasive Vagus Nerve Stimulation (nVNS) on Symptoms and Brain Mechanisms in Premenopausal Women With Temporomandibular Disorders (TMD)
Brief Title: Effects of Vagus Nerve Stimulation on Temporomandibular Disorders.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arpana Church (Other)
Responsible Party: Sponsor-Investigator, Arpana Church, Principal Investigator, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 25-0801
Record Dates: First submitted 2025-12-05; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: TMD; Temporomandibular Disorders (TMDs)
Keywords: TMD; Temporomandibular Disorders; non-invasive vagus nerve stimulation; nVNS
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Pilot/Feasibility, Pre/Post Intervention Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active nVNS Treatment (Experimental): nVNS Treatment 2x/week for 8 weeks
  Interventions: Device: nVNS Treatment

INTERVENTIONS:
Device: nVNS Treatment — nVNS treatment 2x/week for 8 consecutive weeks.
  Other Names: vagus nerve stimulation; non-invasive vagus nerve stimulation

SUMMARY:
The study aims to examine the effects of transcutaneous non-invasive vagus nerve stimulation (nVNS) on symptoms and brain mechanisms in premenopausal women with temporomandibular disorders (TMD). Non-invasive vagus nerve stimulation (nVNS) is the most well researched and possibly the most effective non-invasive neuromodulation treatment for chronic pain conditions that targets the brain-gut-microbiome (BGM) axis.

Participants will be asked to come in for 2 in-clinic visits, at baseline and post treatment. Participants will also be asked to come in 2x/week for 8 consecutive weeks to receive the nVNS treatment. The in-clinic visits will include physical measures, blood draw, saliva sample, and brain MRI. Participants will be asked to collect a stool sample at home and answer online questionnaires regarding, mood, pain, and health behaviors at home, prior to the in-clinic appointments.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50
* Premenopausal menstruating women*
* Participants report or present with at least 1 of 3 cardinal signs of TMD: jaw pain, limited mouth opening, or TMJ noise.
* Specific screening reveals clinical findings that require standard of care medically-indicated intra-articular procedure for management of symptoms including TMJ pain, intra-articular joint disorder leading to joint locking or limited mouth opening or displacement, and severe degenerative joint disease.
* Must have a negative urine test for pregnancy
* Ability to speak the English language fluently due to the standardized assessments involved
* Right-handed (participants are limited to right-handed individuals to reduce variability in brain lateralization and ensure more consistent, interpretable data).

  * Only premenopausal women are included to control for hormonal variability that may influence the results. Participants will be scheduled during their follicular phase based on self-reported last menstrual period to further reduce hormonal confounds.

Exclusion Criteria:

* Medical condition, laboratory finding, or physical exam finding that precludes participation, such as systemic arthritides, juvenile idiopathic arthritis, idiopathic condylar resorption, connective tissue disorders, mandibular osteonecrosis, mandibular and condylar fractures, salivary gland disorders (incl. history of stones or swelling), neoplasms, neurologic/neuropathic, endocrine, or immune/autoimmune diseases and congenital or developmental disorders.
* Pathologic processes found on imaging including neoplasm (Exception: disc displacements and osseous pathology including osteoarthritis/osteoarthrosis).
* Radiation treatment to head and neck
* Prior jaw or open TMJ (including contralateral joint) surgery including plication, chondroplasty, joint replacement, disectomy, and discoplasty.
* Intra-articular therapies of TMJ being sampled that include arthrocentesis, visco-supplementation, and steroid, platelet-rich plasma/platelet-rich fibrin administration within the last 6mo
* Recent febrile illness within the past 8 weeks that precludes or delays participation by more than 90 days
* Trauma to jaw in the last 2mo
* Presence of non-TMD orofacial pain disorders excluding comorbidity of interest (fibromyalgia).
* Pregnancy or lactation
* Undergoing or previously undergone bone anabolic or other hormonal therapies for medical needs
* Unable to participate due to language barrier or mental/intellectual incompetence
* Use of antidepressant drugs unless the participants have been on a stable dose for 60 days.
* Drug and/or alcohol abuse in the past year
* Ongoing dental treatments requiring invasive procedures (e.g. implant placement, tooth extractions, etc.)
* Recent dental treatments within past two weeks that required sustained mouth opening for more than 20 minutes.
* Wearing removable or implant supported dentures or fixed orthodontic appliances
* Unable or unwilling to give informed consent
* Participation in another clinical study that interferes with participation in this study
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.
* Presence of non-TMD orofacial pain disorders such as that from periodontal disease and carious lesions.
* Presence of major psychiatric diagnosis such as schizophrenia, bipolar disorder, post-traumatic stress disorder, obsessive compulsive disorder, or current history of drug or alcohol abuse.
* Individuals with current regular use of narcotics and/or opioids. Use of centrally acting medications that will interfere with neuroimaging testing, such as systemic steroids, opiate analgesics.
* Smokes/Vapes tobacco more than 1/3 pack per day

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | From the baseline in-clinic visit through 8 weeks of biweekly visits, assessed immediately before and after each nVNS session.
  To be measured using a numeric rating scale 0-10.
Pain Unpleasantness | From the baseline in-clinic visit through 8 weeks of biweekly visits, assessed immediately before and after each nVNS session.
  To be measured using a visual analog scale.
Positive and Negative Affect | From the baseline in-clinic visit through 8 weeks of biweekly visits, assessed immediately before and after each nVNS session.
  To be measured using the positive and negative affect scale (PANAS).